CLINICAL TRIAL: NCT07205796
Title: A Phase 2, Randomized, Multicenter, Active-controlled, Double-blind Study to Evaluate the Safety, Reactogenicity, and Immunogenicity of a 2-dose Regimen of Herpes Zoster IN001 mRNA Vaccine (IN001) in Healthy Participants 50 to 79 Years Old
Brief Title: A Phase 2 Study to Describe the Safety, Reactogenicity, and Immunogenicity of Herpes Zoster IN001 mRNA Vaccine (IN001) in Healthy Participants
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shenzhen Shenxin Biotechnology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IN001005
Record Dates: First submitted 2025-09-26; First posted 2025-10-03 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Herpes Zoster
Keywords: IN001; mRNA Vaccine; Vaccine; Varicella-zoster Virus; VZV; Viral Diseases; Shingles; Messenger RNA; Herpes Zoster (HZ); Skin Diseases, Infectious; Safety; Reactogenicity; Immunogenicity; Innorna; Shenxin; Herpesviridae Infections; DNA Virus Infections; Infections; Varicella Zoster Virus Infection; Skin Diseases, Viral; Skin Diseases
MeSH Terms: conditions — Herpes Zoster; Chickenpox; Virus Diseases; Skin Diseases, Infectious; Herpesviridae Infections; DNA Virus Infections; Infections; Varicella Zoster Virus Infection; Skin Diseases, Viral; Skin Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- IN001 Dose A (Arm 1) (Experimental): Participants will receive IN001 at dose level A by IM injection on Day 0 and Day 56.
  Interventions: Biological: HZ Vaccine (IN001)
- IN001 Dose B (Arm 2) (Experimental): Participants will receive IN001 at dose level B by IM injection on Day 0 and Day 56.
  Interventions: Biological: HZ Vaccine (IN001)
- IN001 Dose C (Arm 3) (Experimental): Participants will receive IN001 at dose level C by IM injection on Day 0 and Day 56.
  Interventions: Biological: HZ Vaccine (IN001)
- Shingrix (Arm 4) (Active Comparator): Participants will receive Shingrix by IM injection on Day 0 and Day 56.
  Interventions: Biological: Shingrix

INTERVENTIONS:
Biological: HZ Vaccine (IN001) — Formulation for injection
  Arms: IN001 Dose A (Arm 1); IN001 Dose B (Arm 2); IN001 Dose C (Arm 3)
Biological: Shingrix — Sterile suspension for injection
  Arms: Shingrix (Arm 4)

SUMMARY:
The study will evaluate the safety, tolerability, and immunogenicity (your immune system's reaction) of 3 dose levels of the study vaccine called Herpes Zoster IN001 mRNA Vaccine (IN001) in healthy participants who are between 50 and 79 years of age.

ELIGIBILITY:
Key Inclusion Criteria:

1. Male or female adults, of any race or ethnicity, between 50 and 79 years of age, inclusive, at Screening.
2. Male and female participants must have a body mass index between 18.5 and 34.9 kg/m^2, inclusive, at Screening, and body weight ≥ 50 kg for males and ≥ 45 kg for females.
3. Participants must be able to freely provide documented informed consent prior to study procedures being performed.
4. Participants must be in good general health as determined by comprehensive evaluation by Investigators at the time of enrollment.
5. Participants with asymptomatic medical conditions that are not associated with end-organ damage may be include provided that they are being appropriately treated as per standard of care, are clinically stable, and are not receiving treatments what would be exclusionary in the opinion of the Investigator.
6. Participants must be able and agree to comply with all study visits and procedures (including blood tests, diary completion, receipt of telephone calls from the site, willingness to be available for unscheduled clinic visits).
7. Females of reproductive age will not be pregnant or lactating.
8. Females of childbearing potential, who are sexually active and at risk for pregnancy with their partner(s), must have used appropriate method of contraception at least 30 days prior to enrollment and agree to use a highly effective method of contraception consistently and correctly from enrollment to Study Day 236 (6 months after second vaccination). The Investigator or designee, in consultation with the participant, will confirm that the participant has selected an appropriate method of contraception for the individual participant and his or her partner from the list of appropriate contraception methods and will confirm that the participant has been instructed in its consistent and correct use.
9. Participants must be willing to refrain from blood donation throughout study participation.

Key Exclusion Criteria:

1. Participants with a known history of HZ.
2. Participants with a known history of GBS, encephalomyelitis, or transverse myelitis.
3. Participants with a known history of severe heart disease (i.e., heart failure, recent coronary artery disease, myocarditis, pericarditis, or cardiomyopathy).
4. Participants with acute medical illness or febrile illness, including oral temperature ≥ 38.0°C (≥ 100.4°F) within 1 day prior to Screening. These individuals may be offered the opportunity to enter the study after the fever and/or acute illness has been resolved.
5. Participants with any medical, neurological, or psychiatric condition that, in the opinion of the Investigator, could place the participant at an unacceptable risk of injury or render the participant unable to comply with all study procedures and achieve successful completion of the trial.
6. Participants with a known history of hypersensitivity reactions including anaphylaxis and urticaria, or other significant adverse reactions to IN001 or its excipients; or participants with a known history of severe allergic reaction (e.g., anaphylaxis) to any mRNA vaccine (e.g., COVID-19 mRNA vaccine, RSV mRNA vaccine), any component of SHINGRIX^TM, or after a previous dose of SHINGRIX^TM.
7. Participants who have a positive pregnancy test at the screening visit or who intend to become pregnant during or breastfeed through Study Day 236 (6 months after second vaccination).
8. Participants with uncontrolled hypertension (supine systolic blood pressure [BP] > 140 mmHg or supine average diastolic BP > 90 mmHg at Screening). Eligibility may be reassessed with a single repeat measurement at the Investigator's discretion, and the repeat value will be used for determination.
9. Participants with a history of significant hematologic abnormalities or history of thrombosis with thrombocytopenia syndrome.
10. Participants with hematology and/or clinical chemistry laboratory result(s) that meet the definition of a Grade ≥ 2 abnormality as delineated in the FDA guidance. However, if the institutional normal reference ranges differ from those defined by the region or site, exceptions may be considered on a case-by-case basis with the agreement of the Investigator and the Sponsor.
11. Participants with a history of congenital or acquired immunodeficiency.
12. Participants with an immunosuppressive or immunodeficient state, asplenia, or recurrent severe infections.
13. Participants with a known history of chronic infection of human immunodeficiency virus (HIV), hepatitis B virus (HBV), hepatitis C virus (HCV), or active tuberculosis.
14. Positive HBV and HCV panel and/or positive HIV test. Participants whose results are compatible with prior immunization (indicating evidence of protection) may be included at the discretion of the Investigator that take into account factors such as the timing and effectiveness of the previous immunization.
15. Participants with positive syphilis test.
16. Participants with chronic illness that, in the opinion of the Investigator, is at a stage where it might interfere with trial participation or interpretation of study results.
17. Participants with a known history of vaccination against varicella or HZ.
18. Participants who have received immunoglobulins and/or any blood or blood products within 4 months before the first study vaccination or who plan to receive such products at any time during the study.
19. Participants who have received immunomodulatory, immunostimulatory, or immunosuppressant drugs including interferon and cytotoxic drugs within 3 months of Screening (or 5 half-lives, whichever is longer) or who plan to receive them across the duration of the study.
20. Participants requiring systemic corticosteroids exceeding 10 mg/day of prednisone equivalent for ≥ 10 days within 30 days of Screening. The use of topical, ophthalmic, inhaled, and intranasal steroid preparations will be permitted.
21. Participants who have received or plan to receive any licensed vaccine ≤ 28 days prior to the first vaccination (Day 0) or who plan to receive a licensed vaccine ≤ 28 days after the first study vaccination or ≤ 28 days before or after the second study vaccination. The only exception is licensed inactivated influenza vaccine or non-replicating influenza vaccine, which may be given ≥ 14 days before or ≥ 28 days after receipt the first or second study vaccination.
22. Participants receiving treatment with another investigational drug, biological agent, or device ≤ 28 days of Screening, or 5 half-lives of the investigational drug, whichever is longer; or currently enrolled in or plans to participate in another clinical trial with an investigational agent during the study period (including the follow-up period of the study).
23. Participants with history of drug abuse within 1 year prior to Screening or recreational use of soft drugs (such as marijuana) within 1 month or hard drugs (such as cocaine, phencyclidine, opioid derivatives including heroin, and amphetamine derivatives) within 3 months prior to Screening.
24. History of alcohol abuse within 1 year prior to Screening or regular use of alcohol within 6 months prior to Screening that exceeds 10 units for women or 15 units for men of alcohol per week.
25. Positive alcohol breath test result or positive urine drug screen (UDS) caused by misuse of soft drugs, hard drugs or abuse of any other concomitant medications at Screening and/or on Study Day 0.
26. Participants who are Investigator site staff members, employees of the Sponsor or the clinical research organization directly involved in the conduct of the study, or site staff members otherwise supervised by the Investigator or immediate family members of any of the previously mentioned individuals.
27. Participants with a demonstrated inability to comply with the study procedures.
28. Anything that the Investigator considers would jeopardize the safety of the participant, prevent complete participation in the study, or compromise interpretation of study data.

Ages: 50 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2026-05-01 (Estimated); Primary Completion 2027-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Geometric Mean Concentration (GMC) of Anti-glycoprotein E (gE) Antibodies as Measured by Enzyme-Linked Immunosorbent Assay (ELISA) | Baseline (before first vaccination); 28 days post-second vaccination
Change from Baseline in Geometric Mean Fold Rise (GMFR) of Anti-gE Antibodies as Measured by ELISA | 28 days post-second vaccination
Geometric Mean Titer (GMT) of Anti-VZV Neutralizing Antibodies as Measured by Neutralization Assay | Baseline (before first vaccination); 28 days post-second vaccination
Change from Baseline in GMFR of Anti-VZV Neutralizing Antibodies as Measured by Neutralization Assay | 28 days post-second vaccination
Proportion of Participants with Vaccine Response in Anti-gE Antibodies as Measured by ELISA | 28 days post-second vaccination
Proportion of Participants with Vaccine Response in Anti-VZV Neutralizing Antibodies as Measured by Neutralization Assay | 28 days post-second vaccination
Percentage of Participants Reporting Solicited Local Reactions | For 14 days after each vaccination
Percentage of Participants Reporting Solicited Systemic Events | For 14 days after each vaccination
Percentage of Participants With Unsolicited Adverse Events (AEs) | For 28 days after each vaccination
Percentage of Participants With Any Medically Attended AEs (MAAEs) | From the first vaccination to 6 months after the second vaccination
Percentage of Participants With Any Serious Adverse Events (SAEs), Adverse Events of Special Interest (AESIs), AEs Leading to Vaccine Discontinuation, and AEs Leading to Study Withdrawal | From the first vaccination to 12 months after the second vaccination

SECONDARY OUTCOMES:
GMC of Anti-gE Antibodies as Measured by ELISA | Baseline (before first vaccination); 28 and 56 days post-first vaccination; 14 days and 3, 6 and 12 months post-second vaccination
Change from Baseline in GMFR of Anti-gE Antibodies as Measured by ELISA | 28 and 56 days post-first vaccination; 14 days and 3, 6 and 12 months post-second vaccination
GMT of Anti-VZV Neutralizing Antibodies as Measured by Neutralization Assay | Baseline (before first vaccination); 56 days post-first vaccination; 6 and 12 months post-second vaccination
Change from Baseline in GMFR of Anti-VZV Neutralizing Antibodies as Measured by Neutralization Assay | 56 days post-first vaccination; 6 and 12 months post-second vaccination
Proportion of Participants with Vaccine Response in Anti-gE Antibodies as Measured by ELISA | 28 and 56 days post-first vaccination; 14 days and 3, 6 and 12 months post-second vaccination
Proportion of Participants with Vaccine Response in Anti-VZV Neutralizing Antibodies as Measured by Neutralization Assay | 56 days post-first vaccination; 6 and 12 months post-second vaccination
gE-specific T Cell Response (IFN-γ and IL-4 Secreting T Cells) as Measured by Enzyme-Linked Immunospot (ELISpot) | Baseline (before first vaccination); 28 and 56 days post-first vaccination; 28 days and 3, 6 and 12 months post-second vaccination
Frequencies of gE-specific CD4+ and CD8+ T Cells Expressing Activation Markers (i.e., IFN-γ, IL-2, TNFα, CD40L) as Measured by Intracellular Cytokine Staining (ICS) | Baseline (before first vaccination); 56 days post-first vaccination; 14 and 28 days post-second vaccination

IPD SHARING:
Plan to Share IPD: Undecided